CLINICAL TRIAL: NCT01563848
Title: Cryoablation in Patients With Atrial Flutter
Acronym: CIAFL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAF-712
Record Dates: First submitted 2012-03-23; First posted 2012-03-27 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Atrial Flutter
MeSH Terms: conditions — Atrial Flutter | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (RFA CTI+Reveal) (Active Comparator): assessing the incidence of atrial fibrillation in patients with atrial flutter
  Interventions: Procedure: Implantation of loop recorder; Procedure: Radiofrequency ablation
- Group 2 (RFA CTI+Cryo PVI+Reveal) (Active Comparator): efficacy of cryoablation in patients with atrial flutter
  Interventions: Procedure: Cryoballoon ablation; Procedure: Implantation of loop recorder; Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Cryoballoon ablation — After double transseptal puncture, selective PV angiography was performed to identify the PV ostia in 2 projections (right anterior oblique 30º, left anterior oblique 40 º). Baseline potentials of all PVs were recorded with a Lasso catheter (Biosense Webster, Inc., Diamond Bar, California). To assess the exact position of the inflated balloon in relation to the left atrial (LA)-PV junction, contrast medium was injected from the distal lumen of the cryoballon catheter . CBA was performed for a target time of 300 seconds. The right phrenic nerve was constantly paced from the superior caval vein during freezing at the septal PVs. After each freeze, PV conduction was revaluated by the Lasso catheter.
  Arms: Group 2 (RFA CTI+Cryo PVI+Reveal)
Procedure: Implantation of loop recorder — The RevealXT was implanted in the parasternal area of the chest. The requirement for defining the exact final position was an R-wave amplitude ≥0.4 mV assessed through the Vector Check.
  Patients were provided with the Patient Assistant, a toolthat allows each patient to store the ECG through the implanted device during symptoms: datawere collected in order to analyze heart rhythm during symptomatic events
Procedure: Radiofrequency ablation — Externally-irrigated tip (5-mm tip, Celsius Thermo-Cool, Biosense Webster, Diamond Bar, CA, USA). Temperature-controlled RF delivery was performed with a maximum power output of 50 W and temperature limit of 50 C. The catheter was irrigated using 0.9% saline infusion at a ﬂow rate of 20-40 mL/min during RF delivery and 2 mL/min between applications using a commercially available pump (Cool Flow, Biosense Webster).

SUMMARY:
The investigators hypothesized that revealing the incidence of AF following RFA of the CTI and cryoablation PVI reduces incidence of AF following RFA of the CTI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ECG documented paroxysmal or persistent AFL
* No prior documented history of AF
* Patient undergoing RFA of the CTI for AFL.
* No indication (other than AFL) for continued anticoagulation with warfarin.
* No existing implantable cardiac device (pacemaker, defibrillator, cardiac resynchronization therapy device)
* Availability of an analog phone line.

Exclusion Criteria:

* a history of atrial fibrillation
* Previous AF ablation procedure
* Congestive heart failure
* Left Ventricle ejection fraction less than 35%
* Unwillingness to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-09; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of AF burden | 3 years

SECONDARY OUTCOMES:
All-cause death | 3 years
thromboembolic events | 3 years
hospitalizations | 3 years
procedural complications | 3 years
drug adverse effects | 3 years
number of crossovers | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny A Pokushalov, MD, PhD, Principal Investigator — State Research Institute of Circulation Pathology
Locations (1):
- State Research Institute of Circulation Pathology, Novosibirsk, Russia

REFERENCES:
- [Derived] Romanov A, Pokushalov E, Bayramova S, Ponomarev D, Shabanov V, Losik D, Stenin I, Elesin D, Mikheenko I, Steinberg JS. Prophylactic pulmonary vein isolation during isthmus ablation for atrial flutter: Three-year outcomes of the PREVENT AF I study. J Cardiovasc Electrophysiol. 2018 Jun;29(6):872-878. doi: 10.1111/jce.13485. Epub 2018 Apr 6. PMID 29570894
- See also: State Research Institute of Circulation Pathology Official Site — http://meshalkin.ru